CLINICAL TRIAL: NCT01644994
Title: Phase I Dose-Escalation /Phase II Monocentric Open Trial for Evaluation of Safety and Efficacy of Intracavitary Cisplatin-Fibrin Localized Chemotherapy After Pleurectomy/Decortication or Extrapleural Pneumonectomy for the Treatment of Patients With Malignant Pleural Mesothelioma
Brief Title: Intracavitary Cisplatin-Fibrin Localized Chemotherapy After P/D or EPP for Malignant Pleural Mesothelioma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Swiss National Science Foundation (Other); Swiss Accident Insurance Fund SUVA (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INFLuenCe - Meso
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Malignant Pleural Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant

STUDY DESIGN:
Intervention Model Description: Open Label, single dose local intracavitary application of Cisplatin bound to Fibrin after surgery (removal of Tumor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intracavitary cisplatin-fibrin (Experimental): single dose local intracavitary cisplatin-fibrin application after pleurectomy/decortication
  Interventions: Combination Product: intracavitary cisplatin-fibrin

INTERVENTIONS:
Combination Product: intracavitary cisplatin-fibrin — single dose, local intracavitary application of cisplatin-fibrin after pleurectomy/decortication

SUMMARY:
The aim is to introduce a new therapeutic method of intracavitary chemotherapy (cisplatin) combined with a fibrin carrier (Vivostat®) after pleurectomy/decortication or extrapleural pneumonectomy in a phase I and II study for Malignant Pleural Mesothelioma patients by evaluation of the safety in a dose-escalating model (phase I), and confirmation of safety and efficacy in phase II with the maximum tolerated dose in phase I.

ELIGIBILITY:
Inclusion criteria:

* Patient is able to understand and willing to sign a written informed consent document.
* Male or female, age >=18 years
* ECOG performance status =<2 (ECOG = Eastern Cooperative Oncology Group)
* Resectable MPM (Malignant Pleural Mesothelioma) histologically confirmed (phase I: stage cT1-cT4 cN0-cN3 cM0-cM1 / phase II: stage cT1-cT3 cN0-cN1 cM0) (TNM Tumor staging abbreviations: c = clinical; T = Tumor, N = lymph Nodes, M = Metastases; numbers = quantity)
* Only Phase II: Mediastinal staging (cytological or histological)
* Only Phase II: Induction chemotherapy (3 or more cycles cisplatin or carboplatin (also in combination with other therapeutic agents)
* Patient qualifying for (extended) pleurectomy/decortication ((e)P/D) or extrapleural pneumonectomy (EPP) for resection of MPM, which has to be assessed during a multidisciplinary tumor board including a thoracic surgeon
* Patient must have appropriate organ and bone marrow function as defined: hematologic function: hemoglobin ≥100 g/L, WBC (white blood cell count) ≥3.5 G/L, neutrophils ≥1.5 G/L, thrombocytes ≥100 G/L; liver function: total bilirubin and LDH (lactate dehydrogenase) ≤1.5 x ULN (upper limit of normal); AST (aspartate aminotransferase), ALT (alanine aminotransferase), GGT (gamma glutamyltransferase), and AP (alkaline phosphatase) ≤2.5 x ULN; renal function: creatinine ≤130 μmol/L or, if greater, creatinine clearance ≥60 ml/min/1.73m2.
* Patient must have an appropriate blood coagulation for P/D or EPP (Quick-test > 50%, INR (international normalized ratio) <=1.2)
* The patient agrees to use an efficient contraceptive treatment up to 3 months after cisplatin application if required (pre-menopausal women and men in a sexually mature age).
* Heart and lung function allowing P/D under general anesthesia

Exclusion criteria:

* Known or suspected unwillingness of the patient to follow the rules of the protocol
* Patient who has not recovered from side effects from prior chemotherapy or radiotherapy.
* Any known hypersensitivity against cisplatin or other platinum containing substances or any other components used for the preparation of the drugs.
* Patient must not receive any other investigational agents 4 weeks before treatment and until the end of the observation period (2 months after treatment).
* Patient with prior ipsilateral pleurectomy
* Only Phase II: Multimodality Prognostic Score (MMPS) > 2:

  4 items with a maximum possible score of 4 if the patient presented all four conditions and 0 if none were present: Tumor volume before induction chemotherapy > 500 ml, non-epithelioid histotype in the diagnostic biopsy before induction chemotherapy, CRP (C reactive protein) value > 30 mg/l before induction chemotherapy, and progressive disease after induction chemotherapy according to RECIST criteria
* Patient with uncontrolled intercurrent illnesses that would limit the operative procedure of P/D / EPP or compliance with study requirements
* Tinnitus impairment of more than severity grade I (slight) evaluated by the tinnitus questionnaire MiniTF12_CH (Mini Tinnitus Fragebogen 12, CH = Confoederatio Helvetica (Swiss version)), and/or restricted power of hearing until 4 kHz (kilohertz) confirmed by audiometry, unless age-related presbyacusis in a normal range confirmed by an audiologist.
* Known alcohol and/or drug abuse at the time of screening
* Pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety) | during 6 weeks after surgery with local cisplatin-fibrin application
  (Serious) Adverse Events & safety blood parameters (hematology and clinical chemistry)
Cisplatin concentration in the superficial chest wall tissue | 90 min after application
  local cisplatin concentration in the superficial chest wall biopsy measured by inductively coupled plasma sector field mass spectrometric (ICP-MS) detection

SECONDARY OUTCOMES:
overall survival | up to 5 years (phase I), up to 2 years (phase II)
  time between date of treatment and time point of death or last follow-up, method of Kaplan and Meier
FFR (= Freedom From Recurrence) | 4, 16 weeks, then every 4 months up to 5 (phase I) / 2 years (phase II)
  time to tumor progression by CT or PET-CT/MRI, method of Kaplan and Meier
in-treatment-field FFR (= Freedom From Recurrence) | up to 2 years (phase II)
  time to tumor progression by CT or PET-CT/MRI in the chest cavity where the investigational medicinal product was applied, method of Kaplan and Meier (PET-CT = positron emission computed tomography)
Quality of Life SF-36 (= Short Form-36) | phase I: 0, 4, 8, 16 weeks and every 4w up to 5y; phase II: 0, 6, 16w and every 4w up to 2y
  change from baseline in SF-36 quality of life questionnaire
Quality of Life EORTC QLQ-C15/LC13 (QLQ = Quality of Life Questionnaire, C = Cancer, LC = Lung Cancer) | phase I: 0, 4, 8, 16 weeks and every 4w up to 5y; phase II: 0, 6, 16w and every 4w up to 2y
  change from baseline in EORTC Lung Cancer Questionnaire QLQ-C15/LC13
pharmacokinetics cisplatin concentration in blood serum | baseline, and 0, 2, 6, 10, 24, 48, 120 h postoperative
  cisplatin concentration in blood serum by inductively coupled plasma sector field mass spectrometric (ICP-MS) detection
pharmacokinetics cisplatin concentration in urine | baseline, collection of first 48h, day 14 postoperative
  pharmacokinetics, cisplatin concentration in urine by inductively coupled plasma sector field mass spectrometric (ICP-MS) detection
TUNEL assay | before and 90 min after cisplatin-fibrin application
  markers for apoptosis in superficial chest wall tissue
PAI-1 and p21 (PAI-1 = Plasminogen Activator Inhibitor Typ 1, p21 = CDK-Inhibitor 1 = Cyclin Dependent Kinase Inhibitor 1)) | before and 90 min after cisplatin-fibrin application
  markers for senescence in superficial chest wall tissue

OTHER OUTCOMES:
pharmacokinetics cisplatin concentration in pleural effusion | Pleural effusion collection: 0-48 h postoperative
  cisplatin concentration in pleural effusion by inductively coupled plasma sector field mass spectrometric (ICP-MS) detection

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Opitz, Professor MD, Principal Investigator — University Hospital Zurich, Division of Thoracic Surgery
Locations (1):
- University Hospital Zurich, Division of Thoracic Surgery, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No